CLINICAL TRIAL: NCT06727513
Title: A Two-Operator Technique for GlideScope-Assisted Endotracheal Intubation: Does It Yield a Similar Success Rate? A Randomized Controlled Trial
Brief Title: A Two-Operator Technique for GlideScope-Assisted Endotracheal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Roland Kaddoum, Principal Investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-2024-0231
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication; Airway Trauma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): A single-operator technique for GlideScope intubation.
  Interventions: Procedure: A single-operator technique for GlideScope intubation.
- Experimental (Experimental): A double-operator technique for GlideScope intubation
  Interventions: Procedure: A double-operator technique for GlideScope intubation

INTERVENTIONS:
Procedure: A single-operator technique for GlideScope intubation. — A single-operator technique where the senior resident will insert the GlideScope and perform the endotracheal intubation using an angulated stylet.
  Arms: Control
Procedure: A double-operator technique for GlideScope intubation — A double-operator technique where the senior resident will insert the GlideScope until visualizing an optimal glottic view, then the attending physician will take over the GlideScope keeping it in the same fixed position, while the resident performs the endotracheal intubation using an angulated stylet.
  Arms: Experimental

SUMMARY:
The primary objective of this study is to compare the first attempt success rate of endotracheal intubation using the GlideScope video laryngoscope when performed by two operators versus a single operator.

Secondary objectives include assessing the time to intubate, the need for optimization maneuvers, the effect of the presence of predictors of difficult intubation, the occurrence of adverse events during intubation such as oxyhemoglobin desaturation to less than 90% measured by pulse oximetry, the incidence of airway trauma, and the incidence and severity of post-op sore throat. The main question it aims to answer is: Is endotracheal intubation performed using the Glidescope video laryngoscope with an intubating stylet by two operators, non-inferior to the same procedure performed by single operator in terms of first attempt success rate? Researchers will compare first attempt success rate of endotracheal intubation using the GlideScope video laryngoscope when performed by two operators versus a single operator to see if assistance in using the GlideScope provides similar first attempt success rate of endotracheal intubation and thus guarantees securing a difficult airway.

Participants will be enrolled in one of two groups over 9 months of work. They will be further stratified into blocks according to the presence of at least one predictor of difficult intubation. Patients allocated to the control group will be intubated using the GlideScope by a single operator and those allocated to the experimental group will be intubated using the GlideScope with the assistance of a second operator.

DETAILED DESCRIPTION:
GlideScope-assisted flexible fiberoptic intubation has been successfully used in cases of anticipated and unexpected difficult airways. This technique depends on two operators where the second operator assists in holding the GlideScope while intubation is being attempted by the first operator. However, it is not yet established whether this two-operator technique has any effect on the success rate of first-attempt intubation by the GlideScope video laryngoscope. The primary objective of this study is to compare the first attempt success rate of endotracheal intubation using the GlideScope video laryngoscope when performed by two operators versus a single operator.

Secondary objectives include assessing the time to intubate, the need for optimization maneuvers, the effect of the presence of predictors of difficult intubation, the occurrence of adverse events during intubation such as oxyhemoglobin desaturation to less than 90% measured by pulse oximetry, the incidence of airway trauma, and the incidence and severity of post-operative sore throat. In this prospective randomized controlled trial, 428 patients (214 in each group) adult patients will be enrolled in one of two groups over 9 months of work. They will be further stratified into blocks according to the presence of at least one predictor of difficult intubation. Patients allocated to the control group will be intubated using the GlideScope by a single operator (the resident on the study). Those allocated to the experimental group will be intubated using the GlideScope with the assistance of a second operator (the resident and the attending physician). In both groups, the time to intubate will be measured by the attendings on the study, along with other parameters collected by the resident on the study. If intubation fails, the airway will be subsequently managed using any technique deemed appropriate by the attending anesthesiologist. Data comparing the success rate of endotracheal intubation when a second operator assists in holding the GlideScope is missing. This two-operator technique is essential in the new multimodal airway management involving video-assisted flexible fiberoptic intubation. Our study will determine whether the assistance in using the GlideScope provides similar first attempt success rate of endotracheal intubation and thus guarantees securing a difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* Adult population ≥ 18 years of age
* American Society of Anesthesiologists (ASA) Class I to III
* Elective procedures
* Patients requiring orotracheal intubation with a single-lumen tube under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) IV or V
* Emergency procedures
* Patients who require awake or asleep fiberoptic intubation
* Patients who require nasal intubation
* Patients who require double-lumen endotracheal tube (ETT)
* Patients who are already intubated
* Patients who require rapid sequence induction (uncontrolled Gastroesophageal reflux disease (GERD), hiatal hernia, full stomach)
* Patients with an oropharyngeal/laryngeal pathology (tumor, abscess)
* Patients with maxillary or mandibular fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate of endotracheal intubation | Recorded during the procedure
  First attempt success rate of endotracheal intubation measured by Yes/No

SECONDARY OUTCOMES:
Time to intubate | Recorded during the procedure
  Time to intubate measured in seconds
The need for optimization maneuvers | Recorded during the procedure
  The need for optimization maneuvers measured by Yes/No
Occurrence of adverse events during intubation | Recorded during the procedure
  Occurrence of adverse events during intubation such as oxyhemoglobin desaturation to less than 90% measured by pulse oximetry
The incidence of airway trauma | Recorded during the procedure
  The incidence of airway trauma measured by Yes/No
Incidence and severity of post-operative sore throat | Post-operative sore throat measured one hour after transfer to post anesthesia care unit
  Incidence and severity of post-operative sore throat measured by Yes/No and low pain/high pain

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kaddoum, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No